CLINICAL TRIAL: NCT06928051
Title: Phase 2 Study of S-892216 in Participants Infected With SARS-CoV-2
Brief Title: A Study of S-892216 in Participants With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2314T1621
Record Dates: First submitted 2025-04-09; First posted 2025-04-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: S-892216; Mpro; Main Protease; Nonstructural Protein 5; nsp5; Protease Inhibitor
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- S-892216: Dose 1 (Experimental): Participants will receive S-892216.
  Interventions: Drug: S-892216; Drug: Placebo
- S-892216: Dose 2 (Experimental): Participants will receive S-892216.
  Interventions: Drug: S-892216
- S-892216: Dose 3 (Experimental): Participants will receive S-892216.
  Interventions: Drug: S-892216
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-892216 — S-892216 will be administered orally as a tablet.
  Arms: S-892216: Dose 1; S-892216: Dose 2; S-892216: Dose 3
Drug: Placebo — Placebo will be administered orally as a tablet.
  Arms: Placebo; S-892216: Dose 1

SUMMARY:
The primary objective of this study is to investigate the antiviral effect of S-892216 in participants with coronavirus disease 2019 (COVID-19) due to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Must weigh ≥40 kilograms
* Must have at least 2 COVID-19 signs/symptoms of mild or higher severity, or at least 1 sign/symptom of moderate or higher severity, within the 72 hours prior to randomization, and the symptoms must still be present in the 24 hours prior to randomization
* Documentation of laboratory-confirmed active SARS-CoV-2 infection, as determined by a nucleic acid (for example, qRT-PCR) or antigen test from any respiratory tract specimen (for example, oropharyngeal, NP or nasal swab, or saliva), or any other SARS-CoV-2 test approved according to local regulations, collected ≤72 hours (3 days) prior to randomization
* Oxygen saturation (SpO2) of ≥92% on room air adjusted for altitude and obtained at rest by study staff within the 24 hours prior to randomization. For a potential participant who regularly receives chronic supplementary oxygen for an underlying lung condition, SpO2 measured while on standard home oxygen supplementation level must be ≥92%.
* Capable and willing to complete an electronic participant diary
* Contraceptive use by female participants should be consistent with local regulations regarding the use of contraceptive methods for those participating in clinical studies. Note: The investigational medication may lead to an increase or decrease of sex hormone levels; therefore, hormonal contraception must not be used alone and must be combined with a barrier method.
* A woman of childbearing potential must have a negative urine pregnancy test within the 24 hours before the first dose of investigational intervention
* Must be randomized ≤72 hours from onset of COVID-19 symptoms (defined as the time point when at least 1 of the COVID-19 symptoms occurs)
* Agrees to not participate in another clinical trial for the treatment of COVID-19 or SARS-CoV-2 during the study period unless meeting hospitalization criteria or reaching Day 28, whichever is earliest

Key Exclusion Criteria:

* High risk of progression to severe COVID-19, as defined in the protocol
* Documented respiratory infection (for example, influenza, respiratory syncytial virus) other than COVID-19 within the 14 days prior to the screening visit
* Known current renal impairment deﬁned as estimated glomerular filtration rate <60 milliliters/minute/1.73 meters squared or requiring dialysis
* Known history of cirrhosis or liver decompensation (including ascites, variceal bleeding, or hepatic encephalopathy)
* Known history of any of the following abnormalities in the following clinical laboratory tests (within the 6 months prior to the screening visit):

  * Total bilirubin ≥2 × upper limit of normal (ULN) (except for Gilbert's syndrome)
  * Aspartate aminotransferase or alanine aminotransferase ≥2 × ULN
* A QT interval corrected using Fridericia's formula at the screening visit:

  * For males: >450 milliseconds (msec)
  * For females: >470 msec
* History of hospitalization for the current SARS-CoV-2 infection or anticipated need for hospitalization within 24 hours after randomization
* History of cancer except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Women with a history of osteoporosis
* Received or expected to receive any dose of a SARS-CoV-2 vaccine within 14 days of randomization or during the study through day 28
* Received or expected to receive any other COVID-19-specific treatment, including outpatient remdesivir, Paxlovid, molnupiravir, monoclonal antibodies, ensitrelvir, and convalescent plasma for the current COVID-19 infection
* Exposed to an investigational drug within 30 days or 5 half-lives of the drug prior to the screening visit

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 282 (Actual)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in SARS-CoV-2 Viral RNA Level on Day 4 as Assessed by Quantitative Reverse-transcription Polymerase Chain Reaction (qRT-PCR) of Nasopharyngeal (NP) Swabs | Baseline through Day 4

SECONDARY OUTCOMES:
Time to the First Negative SARS CoV-2 Viral RNA qRT-PCR Result | Baseline through Day 28
Time to the First SARS CoV-2 Viral RNA Viral RNA Level Less Than the Lower Limit of Quantitation (LLOQ) | Baseline through Day 28
Number of Participants With a Positive SARS CoV-2 Viral RNA qRT-PCR Test | Baseline, Days 2, 4, 6, 10, 14, 21, and 28
Change From Baseline in SARS CoV-2 Viral RNA Level | Baseline, Days 2, 6, 10, 14, 21, and 28
Area Under the Curve of Change From Baseline in SARS-CoV-2 Viral RNA Level Through Day 4 and Day 6 | Baseline through Day 4 and Day 6
Time to Sustained (2 Consecutive Days) Resolution of COVID-19 Symptoms | Baseline through Day 28
Time to First Resolution of COVID-19 Symptoms | Baseline through Day 28
Time to Return to Pre-COVID-19 Health | Baseline through Day 28
Plasma Concentration of S-892216 | Days 2, 6, and 10

CONTACTS AND LOCATIONS:
Locations (57):
- United States (21):
  - Healthstar Research, Hot Springs, Arkansas
  - Invictus Clinical Research Group LLC, Coconut Creek, Florida
  - Hope Clinical Trials, Coral Gables, Florida
  - Advanced Research for Health Improvement LLC, Immokalee, Florida
  - LCC Medical Research, Miami, Florida
  - CCM Clinical Research Group, Miami, Florida
  - Global Health Clinical Trials, Miami, Florida
  - Continental Clinical Research, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Kendall South Medical Center Inc, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Quality Research of South Florida, Miami Lakes, Florida
  - Oceane7 Medical & Research Center, Inc., Miami Lakes, Florida
  - Combined Research Orlando Phase I-IV LLC, Orlando, Florida
  - Global Clinical Professionals, St. Petersburg, Florida
  - Balanced Life Health Care Solutions, Lawrenceville, Georgia
  - PanAmerican Clincal Research, Brownsville, Texas
  - Alina Clinical Trials LLC, Dallas, Texas
  - Care United Research, LLC, Forney, Texas
  - Clinical Research Partners LLC, Richmond, Virginia
  - Frontier Clinical Research LLC, Kingwood, West Virginia
- Japan (36):
  - Japanese Site 10, Multiple Locations
  - Japanese Site 11, Multiple Locations
  - Japanese Site 12, Multiple Locations
  - Japanese Site 13, Multiple Locations
  - Japanese Site 14, Multiple Locations
  - Japanese Site 15, Multiple Locations
  - Japanese Site 16, Multiple Locations
  - Japanese Site 17, Multiple Locations
  - Japanese Site 18, Multiple Locations
  - Japanese Site 19, Multiple Locations
  - Japanese Site 1, Multiple Locations
  - Japanese Site 20, Multiple Locations
  - Japanese Site 21, Multiple Locations
  - Japanese Site 22, Multiple Locations
  - Japanese Site 23, Multiple Locations
  - Japanese Site 24, Multiple Locations
  - Japanese Site 25, Multiple Locations
  - Japanese Site 26, Multiple Locations
  - Japanese Site 27, Multiple Locations
  - Japanese Site 28, Multiple Locations
  - Japanese Site 29, Multiple Locations
  - Japanese Site 2, Multiple Locations
  - Japanese Site 30, Multiple Locations
  - Japanese Site 31, Multiple Locations
  - Japanese Site 32, Multiple Locations
  - Japanese Site 33, Multiple Locations
  - Japanese Site 34, Multiple Locations
  - Japanese Site 35, Multiple Locations
  - Japanese Site 36, Multiple Locations
  - Japanese Site 3, Multiple Locations
  - Japanese Site 4, Multiple Locations
  - Japanese Site 5, Multiple Locations
  - Japanese Site 6, Multiple Locations
  - Japanese Site 7, Multiple Locations
  - Japanese Site 8, Multiple Locations
  - Japanese Site 9, Multiple Locations

IPD SHARING:
Plan to Share IPD: No